CLINICAL TRIAL: NCT03682159
Title: The Effect of Manual Lymphatic Drainage on Swelling After Orthognathic Surgery - a Qualitative and 3D Facial Analysis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Tandheelkunde, Prof. Dr. Guy De Pauw, University Hospital, Ghent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: B670201629310
Record Dates: First submitted 2018-09-12; First posted 2018-09-24 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Care/Methods; Drainage/Methods; Edema/Prevention & Control; Orthognathic Surgical Procedures/Adverse Effects
MeSH Terms: conditions — Edema | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention)
- intervention (Experimental)
  Interventions: Other: manual lymphatic drainage

INTERVENTIONS:
Other: manual lymphatic drainage — The intervention group received the same conventional postoperative cares as the control group, but also underwent 5 sessions of manual lymphatic drainage (MLD)
  Arms: intervention

SUMMARY:
Introduction / background

Orthognathic surgery is an operation in which one or both jaws are fixed in a more favorable position performed by an osteotomy. In this way, large skeletal differences between the upper and lower jaw can be corrected surgically. The aim is to obtain a good and stable occlusion as well as to improve the facial aesthetics off the patient, where this would not be possible without surgery. These surgical procedures are accompanied by swelling of the face that can last for several days. The swelling is often considered unpleasant by the patients. The post-operative application of ice on the face can reduce the swelling. Also, performing manual lymphatic drainage (MLD) at the head and neck region would have a positive effect on the swelling after the operation. Manual lymphatic drainage is a kind of gentle massage performed by physiotherapists to reduce swelling in a faster way after surgery. This therapy is performed during the first days after the surgery and lasts about 30 minutes per session. There is still insufficient evidence to be whether or not this technique offers added value for patients undergoing jaw surgery.

Goal

The aim of this study is to investigate whether or not manual lymphatic drainage provides added value for patients undergoing jaw surgery. The facial swelling will be studied as the primary outcome variable. Other postoperative discomforts associated with orthognathic surgery are the secondary outcome variables. This study may or may not justify performing MLD and ensure that it is included in a postoperative protocol.

Methodological approach

The investigators would like to measure and compare the swelling in the face in an objective way between patients who received manual lymphatic drainage (intervention group) and patients who did not undergo manual lymphatic drainage (control group) The control group receives the standard postoperative care that is applied at the University Hospital Ghent. The intervention group also receives the same postoperative cares, as well as 5 MLD sessions during the first postoperative week (1st, 2nd, 3rd, 4th, 7th postoperative day).The objective measurement of the swelling can be done on the basis of a laser scan that can create 3D images of the face. For this, the patient should take a natural head position at rest and have a relaxed facial expression. This technique of imaging is non-invasive and there is no x-ray radiation involved! The 3D images are taken at the following times: 3 days, 1 week, 2 weeks, 1 month, 3 months and 6 months after the operation. Together with the scans, the patients were asked to fill in a questionnaire to frame the subjective postoperative discomfort associated with orthognathic surgery.

The change in swelling can be analyzed on the basis of specific measurements on the 3D images as well as by recording surface changes. The last 3D image is used as a reference to superimpose the other 3D images as there is no longer any swelling on this 3D image. After analyzing these data, it can be assessed to what extent manual lymphatic drainage offers an advantage to reduce swelling after orthognathic surgery.

DETAILED DESCRIPTION:
Subjects

The patients were collected from the maxillofacial department of the University Hospital of Ghent, Belgium between January 2015 and March 2018. The subjects had to meet certain inclusion criteria to participate in this study and they were rejected if one of the mentioned exclusion criteria was presented.

Inclusion criteria:

1. Age 14 - 65 years
2. ASA score I
3. BSSO, LeFort I or Bimax

Exclusion criteria:

1. Transgender patients
2. Other facial surgery's
3. Deviant medication
4. Cleft patients
5. Lot of facial hair
6. Refused to participate

Next, patients who met all inclusion criteria and didn't drop out because of the exclusion criteria, were randomized in 2 treatment groups by block randomization. One group received the conventional postoperative cares from the University Hospital Ghent including topical ice application (also called cryotherapy), standardized medication and postoperative instructions. These patients were used as controls. The other group received the same conventional postoperative cares as mentioned in the control group, but also underwent 5 sessions of MLD after the operation. Starting on the 1st postoperative day. These patients belonged to the intervention group.

Protocol

For every postoperative visit there was a fixed flowchart that needed to be followed. First the patient was asked to fill in the survey which questioned the pain and swelling. When this was done, a 3D face scan was taken of the untouched face in a natural resting position with a laser scanner (Planmeca Proface®, Planmeca Oy, Finland). Thereafter, only the intervention group received a MLD session if indicated by the protocol. Finally, the appointments for the future were checked in order to prevent no-shows. The last visit of every patient was planned 6 months after surgery.

Ethical approval

The study was submitted to the research ethics board of the University Hospital of Ghent and a positive advise was given for this protocol. The study has also been registered (no. B670201629310). A written informed consent was obtained from each subject after the researcher explained the purpose and the procedure of the study containing the possible risks and benefits associated with the interventions.

Manual Lymph drainage

The MLD sessions were performed by 3 masters in physiotherapy (5th years) who were specially calibrated for this study by the same experienced MLD instructor and physiotherapist (V.V.B.). The used method for MLD was these described by Dr. Vodder and is a rather soft kind of massage that lasts for about 40 minutes per session. All MLD session were performed in a pleasant temperature and in an extremely relaxed atmosphere. In order to achieve this, it was requested not to talk during treatment. Also all patients were in a comfortable lying position when the MLD was performed.

Questionnaire

Before taking the face scans, a questionnaire was always filled out by the patient. These questionnaires were created with the aim to give an idea of the perceived swelling and pain. At the end, six questionnaires were collected per patient as prescribed by the protocol.

Pain scores were assessed using a visual analogue scale (VAS) of 100 mm, representing all pain sensations from none to maximum. Zero mm indicates no pain, 50 mm moderate pain and 100 mm worst pain possible. Patients were asked to place a mark along the line that corresponded to the amount of pain they were experiencing. In this questionnaire, two visual analogue scales were used to question the average pain of the last 24 hours and the worst pain of the last 24 hours.

To measure the swelling in an subjective way, a five-point Likert-type scale was used. The patients were asked whether they suffered from swelling in the last 24 hours. Five possible answers could be checked: none, almost none, moderate, pretty much and very much.

Face scan and processing

Six face scans were taken from each patient with the Planmeca Proface® (Planmeca Oy, Finland) as indicated by the protocol. This technique of imaging is non-invasive and there is no x-ray radiation involved! The face scans were transformed into STL files and subsequently exported to software programs.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 - 65 years
* ASA score I
* BSSO, LeFort I or Bimax

Exclusion Criteria:

* Transgender patients
* Other facial surgery's
* Deviant medication
* Cleft patients
* Lot of facial hair
* Refused to participate

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-09; Primary Completion 2018-04 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change of swelling after orthognathic surgery assessed by 3D face scans | At the 3th, 7th and 14th day after surgery, as well as 1 month, 3 months and 6 months after surgery.
  3D face scans were taken with the Planmeca Proface® (Planmeca Oy, Finland) at 6 fixed time points after surgery to measure change in facial swelling. This was done by superimposition of the different scans. Swelling was expressed in millimeters.

SECONDARY OUTCOMES:
Questionnaire with a 100 millimeter Visual Analogue Scale to measure perceived pain | At the 3th, 7th and 14th day after surgery, as well as 1 month, 3 months and 6 months after surgery.
  Pain scores were assessed at 6 fixed time points after surgery using a visual analogue scale (VAS) of 100 mm, representing all pain sensations from none to maximum. Zero mm indicates no pain, 50 mm moderate pain and 100 mm worst pain possible. Patients were asked to place a mark along the line that corresponded to the amount of pain they were experiencing.
Questionnaire with a five-point Likert-type Scale to measure perceived swelling | at the 3th, 7th and 14th day after surgery, as well as 1 month, 3 months and 6 months after surgery.
  Swelling was assessed at 6 fixed time points after surgery using a five-point Likert-type Scale. Five possible answers could be checked: no swelling, almost no swelling, moderate swelling, pretty much swelling and very much swelling.

CONTACTS AND LOCATIONS:
Overall Officials: Guy De Pauw, Prof. Dr., Principal Investigator — University Ghent
Locations (1):
- University of Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yaedu RYF, Mello MAB, Tucunduva RA, da Silveira JSZ, Takahashi MPMS, Valente ACB. Postoperative Orthognathic Surgery Edema Assessment With and Without Manual Lymphatic Drainage. J Craniofac Surg. 2017 Oct;28(7):1816-1820. doi: 10.1097/SCS.0000000000003850. PMID 28872503
- [Background] Szolnoky G, Szendi-Horvath K, Seres L, Boda K, Kemeny L. Manual lymph drainage efficiently reduces postoperative facial swelling and discomfort after removal of impacted third molars. Lymphology. 2007 Sep;40(3):138-42. PMID 18062616